CLINICAL TRIAL: NCT01562262
Title: Behavior of Psychomotor Vigilance Task Performance in Subjects With Obstructive Sleep Apnea With and Without Complaints of Daytime Sleepiness
Brief Title: Comparison of RT in Patients With Sleep Apnea With and Without Complaints of Daytime Sleepiness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Marco Tulio de Mello, PhD Professor, Federal University of São Paulo
Other Study IDs: CEP1122/11
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Sleep Apnea
Keywords: Apnea; PVT; Reaction Time
MeSH Terms: conditions — Sleep Apnea Syndromes; Apnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- CTR: Control group
- ASS: Apnea without complaints group
- ACS: SAOS Group

SUMMARY:
Not all patients with the Obstructive Sleep Apnea Syndrome (OSAS), mostly mild, have excessive daytime sleepiness. Sleep fragmentation provides the performance decrease with increasing reaction time to external stimuli and correlates with excessive sleepiness. So, the study aims at assessing the effect of sleep fragmentation on the Reaction Time and it's maintenance in patients with OSAS compared with healthy, to better clarify were patients with and without somnolence differ. For that, will be recruited 30 male volunteers aged between 20 and 50 year old to participate in the study. They will be distributed in three groups: "CONTROL" (without symptoms of sleepiness and apnea and hypopnea index (AHI) less than 5), "SS" (with AHI between 5 and 15 without symptoms of somnolence) and group "CS" (with AHI between 5 and 15 with symptoms of somnolence). The groups will undergo a polysomnography and subsequently, the Test and Maintenance of Wakefulness and PVT Battery Tests. The reaction time will be compared, as well as the ability to keep the reaction time over time between groups to see whether there is a difference between the motor performance throughout the day and the perception of sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Man
* Aged between 20 and 45 years old
* BMI between 20-30

Exclusion Criteria:

* Cigarette Smoke
* Drug intake
* Other sleep disturbances

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Man, ages between 20 and 45 years with and without drowsiness and no sleep disturbances checked before the study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil